CLINICAL TRIAL: NCT02661100
Title: A Phase I/II Trial of CDX-1401 (a Vaccine Consisting of a Human Monoclonal Antibody Specific for DEC-205, Fused to Full-length Tumor Antigen NY-ESO-1) in Combination With Poly-ICLC and Pembrolizumab, in Previously Treated Advanced Solid Tumor Patients
Brief Title: A Trial of CDX-1401 in Combination With Poly-ICLC and Pembrolizumab, in Previously Treated Advanced Solid Tumor Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Drug unavailable
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2Y16
Record Dates: First submitted 2016-01-19; First posted 2016-01-22 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Non Small Cell Lung Cancer; Advanced Triple Negative Breast Cancer; Small Cell Lung Cancer; Urothelial Cancer; Mesothelioma; Malignant Melanoma
Keywords: Vaccine; NY-ESO-1; DEC-205; Poly-ICLC; Pembrolizumab; Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Mesothelioma; Melanoma; Neoplasms | interventions — pembrolizumab; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CDX-1401 + Poly-ICLC + Pembrolizumab followed by Pembrolizumab (Experimental): Patients receive CDX-1401, Poly-ICLC and Pembrolizumab for 4 cycles (Q 3 weeks) followed by Pembrolizumab alone (Q 3 weeks) until disease progression.
  Interventions: Drug: Pembrolizumab; Biological: CDX-1401; Biological: Poly-ICLC

INTERVENTIONS:
Drug: Pembrolizumab — 200mg/kg by IV infusion on Day 1 of each 3 week cycle. Given until disease progression
Biological: CDX-1401 — 1mg given subcutaneously on day 1 of each 3 week cycle. Given for 4 cycles
Biological: Poly-ICLC — 2mg given subcutaneously on day 1 and 2 of each 3 week cycle. Given for 4 cycles

SUMMARY:
This study will look at the safety of the combination of three drugs (CDX-1401, Poly-ICL, and Pembrolizumab) and its effect on decreasing tumors. Pembrolizumab is an experimental cancer drug. CDX-1401 is a tumor specific antigen and Poly-ICL is a Toll-like receptor agonist tumor specific antigens which when combined with Pembrolizumab may increase the tumor response to this drug.

DETAILED DESCRIPTION:
Antigen presentation and cellular immunity are complex processes, and subject to modulation because of the tumor microenvironment. Antigen presenting cells in the tumor microenvironment acquire the antigens from tumor cells. Tumors express several tumor specific antigens that can be leveraged by the immune system to mount an effective anti-tumor response. NY-ESO-1, one of the cancer testis antigens, is expressed in several tumors including non-small cell lung cancer (NSCLC), triple negative breast cancer (TNBC), and melanoma. NY-ESO-1 is highly immunogenic and spontaneous tumor regressions in association with humoral and cellular responses to NY-ESO-1 have been reported. NY-ESO-1 is tumor specific and is not detected in non-malignant tissues with the exception of germ cells and trophoblasts, thus making it an attractive target for cancer vaccine development. Cancer vaccines can augment the process of cancer specific antigen presentation, however the efficacy of protein-based vaccines is limited due to weak immunogenicity and inefficient uptake by antigen presenting cells for presentation to T and B cells, and lack of targeting to appropriate antigen presenting cells. Dendritic cells (DCs) are highly specialized antigen-presenting cells that play a central role in initiating and regulating immunity. Deca-lectin, DEC-205 (CD205) is a surface receptor of DCs, which is highly expressed by human DCs and can mediate antigen uptake, processing, and presentation. CDX-1401 is a fully human anti-DEC-205 mAb (3G9) genetically fused to the full length NY-ESO-1. In preclinical studies, Dec-205 fused to NY-ESO-was more efficiently cross-presented to T-cells than NY-ESO-1 protein alone. In a recently concluded phase 1 study of CDX-1401 in combination with adjuvant Toll-like receptor agonists with Resiquimod (TLR7/8 agonist) and Hiltonol (poly-ICLC; TLR3 agonist), CDX-1401 was well tolerated with no dose-limiting toxicities and no treatment related grade 3/4 toxicities. Clinical activity was noted in solid tumors including NSCLC. Interestingly, few of the patients who progressed on CDX-1401 subsequently received immune checkpoint inhibitors and several of these patients with NY-ESO-1-specific cellular response had partial responses by RECISTimmune-related response criteria (IRRC). Previous studies reported enhanced T-cell responses in autologous dendritic cell/myeloma fusion vaccines with PD-1 blockade using CT-011 (Anti-PD1 antibody). In addition, increased tumor-infiltrating dendritic cells which are PD1 positive mediate immune suppression and PD-1 blockade in mice ovarian cancer models enhance effector T-cell responses and reduce tumor burden. Thus, we hypothesize that the ability of CDX-1401 to generate an effective anti-tumor immune response could be enhanced when co-administered with an anti-PD1 antibody.

In this study, investigators will examine the safety of the three drug combination of CDX-1401, Poly-ICL (TLR-3 agonist), and Pembrolizumab, and its impact in generating robust and effective anti-tumor immune responses. The preliminary clinical data from Pembrolizumab are promising, and strategies such as this to enhance tumor specific antigen presentation may augment the responses and clinical benefit from Pembrolizumab.

Primary Objective:

To assess the safety, and tolerability of CDX-1401 in combination with Pembrolizumab

Secondary Objectives:

1. To determine whether the anti-tumor response is substantially increased by vaccination with CDX-1401 (anti-DEC205-NY-ESO-1 fusion protein vaccine) in combination with an immune-checkpoint inhibitor, Pembrolizumab (anti-PD1 mAb) in previously treated patients with advanced solid tumors.
2. To determine immune response to NY-ESO-1 and other tumor specific antigens in patients treated with CDX-1401 and Pembrolizumab.
3. To evaluate changes in Tumor infiltrating lymphocytes and other immune evasive pathway biomarkers post treatment with CDX-1401 and Pembrolizumab.
4. To perform exploratory analysis to identify biomarkers to predict both antigen specific T-cell responses and clinical benefit to CDX-1401 and Pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Patients with previously treated advanced lung cancer (NSCLC, SCLC and mesothelioma), advanced triple negative breast cancer, urothelial cancers and malignant melanoma. Tumors should be positive for expression of NY-ESO-1, as assessed by external central laboratory testing.
* Malignancy that has progressed after any therapies with curative potential or at least one approved palliative therapy for which the patient is a candidate. Patients with metastatic melanoma may be enrolled without prior treatment provided they meet rest of the eligibility criteria.
* Where applicable, chemotherapy or radiation therapy must have been completed at least 4 weeks prior to the first dose of study treatment; the interval for prior anticancer therapeutic radiopharmaceuticals is at least 8 weeks. For patients on small molecule tyrosine kinase inhibitors therapy must have been completed 14 days prior to start of study treatment. The patient must have adequately recovered from any clinically significant toxicity experienced during prior treatment(s) in the investigator's opinion.
* Chemoembolization, surgery or any other local therapy completed at least 4 weeks prior to the first dose of study treatment.
* Have measurable disease based on immune-related Response Criteria (irRC).
* Availability of tumor tissue (preferably from a recent biopsy or resection, or if not available, on the archived tumor tissue from the primary resection) for NY-ESO-1 expression analysis. Positive NY-ESO-1 expression will be required for entry. NY-ESO-1 expression will be analyzed at a central laboratory.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* 10. Demonstrate adequate organ function as defined below , all screening labs should be performed within 10 days of treatment initiation.

  * Absolute neutrophil count (ANC) >=1,500/mcL
  * Platelets >= 100,00/mcL
  * Hemoglobin >= 9g/dL or >= 5.6mmol/L without transfusion or EPO dependency (within 7 days of assessment)
  * Serum creatinine =< 1.5X upper limit of normal
  * Measured creatinine clearance >=mL/min for subject with creatinine levels >1.5 X institutional upper limit of normal
  * Serum total bilirubin =< 1.5X upper limit of normal
  * AST (SGOT) =< 2.5 X upper limit of normal or =< 5X upper limit of normal for subjects with liver metastases
  * ALT (SGPT) =< 2.5 X upper limit of normal or =< 5X upper limit of normal for subjects with liver metastases
  * Albumin >= 2.5mg/dL
  * International Normalized Ratio =< 1.5 X upper limit of normal unless subject is receiving anticoagulant therapy as long as Prothrombin Time or Partial Thromboplastin Time is within therapeutic range of intended use of anticoagulants Activated Partial Thromboplastin Time (aPTT) =< 1.5 X upper limit of normal unless subject is receiving anticoagulant therapy as long as Prothrombin Time or Partial Thromboplastin Time is within therapeutic range of intended use of anticoagulants
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential must be willing to use an adequate method of contraception - Contraception, for the course of the study through 120 days after the last dose of study medication.
* Male subjects of childbearing potential must agree to use an adequate method of contraception - Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active bacillus tuberculosis
* Hypersensitivity to Pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody within 4 weeks prior to study day 1 or who has not recovered (ie =< Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (ie =< Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Has a known additional malignancy that is progressing or required active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided therapy are stable (without evidence of progression by imagining for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (ie with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not the best interest of the subject to participate, in the opinion of the treating investigator.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2 agent and previous administration of vaccine therapy targeting NY-ESO-1.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. -- Note: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | Up to 28 days of therapy (Cycle 1)
  Dose limiting toxicity (DLT) will be defined as any side effects which are attributable to the study treatment during the first 28 days of therapy (Cycle 1). The dose limiting toxicity will be based on the tolerability observed during treatment.

SECONDARY OUTCOMES:
Objective Response Rate for combination therapy | Up to 24 months after beginning treatment
  Tumor response will be assessed using immune-related Response Criteria (irRC). The objective response rate will be estimated based on the crude proportion of patients who achieve complete response (CR) or partial response (PR). Complete response is defined as the disappearance of all lesions in two consecutive observations not less than 4 weeks apart. Partial response is defined as >=50% decrease in tumor burden compared with baseline in two observations at least 4 weeks apart.
Median Duration of Response | Up to 24 months after beginning treatment
  Tumor response will be assessed using immune-related Response Criteria (irRC). The duration of response will be calculated from the time when the criteria for response are first met to the first documentation of relapse (after CR) or progression (after PR). Complete response is defined as the disappearance of all lesions in two consecutive observations not less than 4 weeks apart. Partial response is defined as >=50% decrease in tumor burden compared with baseline in two observations at least 4 weeks apart. Stable disease is when 50% decrease in tumor burden compared with baseline cannot be established nor 25% increase compared with baseline. Progressive disease is defined as at least 25% increase in tumor burden compared with baseline in two consecutive observations at least 4 weeks apart.
Median time to tumor response | Up to 24 months after beginning treatment
  Tumor response will be assessed using immune-related Response Criteria (irRC). Complete response is defined as the disappearance of all lesions in two consecutive observations not less than 4 weeks apart. Partial response is defined as >=50% decrease in tumor burden compared with baseline in two observations at least 4 weeks apart. Stable disease is when 50% decrease in tumor burden compared with baseline cannot be established nor 25% increase compared with baseline. Progressive disease is defined as at least 25% increase in tumor burden compared with baseline in two consecutive observations at least 4 weeks apart.
Median time of progression free survival | Up to 24 months after beginning treatment
  Time from beginning of treatment to disease progression. Progressive disease is defined as at least 25% increase in tumor burden compared with baseline in two consecutive observations at least 4 weeks apart.
Median Overall Survival | Up to 24 months after beginning treatment
  Defined as time from beginning of treatment until death, withdrawal of consent, or the end of the study, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Vamsidhar Velcheti, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center